CLINICAL TRIAL: NCT03960541
Title: CD24Fc Administration to Decrease LDL and Inflammation in HIV Patients, Both as Markers of Efficacy and Cardiovascular Risk Reduction (CALIBER)
Brief Title: Efprezimod Alfa (CD24Fc, MK-7110) Administration to Decrease Low-Density Lipoprotein (LDL) and Inflammation in Human Immunodeficiency Virus (HIV) Patients (CALIBER) (MK-7110-003)
Acronym: CALIBER
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Oncoimmune, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7110-003; CD24Fc-003 (Other: OncoImmune, Inc.); HP-00086029 (Other: OncoImmune, Inc.); MK-7110-003 (Other: Merck)
Record Dates: First submitted 2019-05-15; First posted 2019-05-23 (Actual); Results first posted 2022-06-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: HIV Infections; Dyslipidemias
Keywords: HIV Dyslipidemias; CD24Fc; HIV Chronic Inflammation; LDL Reduction
MeSH Terms: conditions — HIV Infections; Dyslipidemias | interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized, double blinded, placebo controlled.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Efprezimod alfa Treatment (Experimental): Participants received an intravenous infusion of 240 mg of efprezimod alfa on Days 0, 14, and 28.
  Interventions: Drug: Efprezimod alfa (human CD24 extracellular domain and human IgG1 Fc fusion protein)
- Placebo (Placebo Comparator): Participants received an intravenous infusion of placebo (sterile saline solution) on Days 0, 14, and 28.
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Efprezimod alfa (human CD24 extracellular domain and human IgG1 Fc fusion protein) — Efprezimod alfa will be given as IV infusion, 240 mg per infusion, on Days 0, 14, and 28.
  Other Names: CD24Fc; MK-7110
  Arms: Efprezimod alfa Treatment
Drug: Saline Solution — Sterile saline solution (0.9% sodium chloride) will be given as placebo via IV infusion, 100 ml per infusion, on Days 0, 14, and 28.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This is a phase 2, randomized, double-blinded, placebo-controlled clinical trial. The intervention drug will be efprezimod alfa (intravenous [IV] infusion). A cohort of 64 patients with HIV on antiretroviral therapy (ART) will be randomized in a 1:1 fashion to be administered 3 doses of efprezimod alfa (240mg IV infusion) or placebo once every 2 weeks (q2w) during a 4-week window, followed by a 24-week follow-up window to assess the changes in LDL.

DETAILED DESCRIPTION:
This study is a phase 2, randomized, placebo-control, double-blinded clinical trial to assess the effect of efprezimod alfa on reduction in low-density lipoprotein (LDL) among patients with HIV. The effect of efprezimod alfa on total cholesterol and triglycerides, markers of immune activation (T cell activation, sCD14, and inflammatory cytokines), size of HIV reservoirs, hemoglobin (HbA1c) and leptin, and hepatic steatosis will be evaluated.

It is hypothesized that therapy with efprezimod alfa will result in significant decreases in LDL in HIV patients. In addition, efprezimod alfa may reduce leptin and cholesterol, HbA1c, hepatic steatosis and fibrosis, and markers of inflammation in patients with chronic HIV who are virally suppressed on ART.

In this phase 2 study, a cohort of 64 HIV patients virally suppressed on ART will be randomized in a 1:1 fashion to receive an intravenous infusion of 240 mg of efprezimod alfa vs. placebo administered every 2 weeks during a 4-week treatment window, followed by a 24- week follow-up period. Patients will be followed for safety and adverse events as well as changes in lipid metabolism and inflammatory markers during a 24-week follow-up period. This investigation will take place at the University of Maryland.

ELIGIBILITY:
Inclusion Criteria:

* Provides signed and dated informed consent form
* Is willing to comply with all study procedures and availability for the duration of the study
* Is at least 50 years of age or older at screening
* Has LDL-C > 70 mg/dL.
* Has a median American College of Cardiology (ACC)/American Heart Association (AHA) atherosclerotic cardiovascular disease (ASCVD) ACC/AHA ASCVD risk score ≥ 7.5%.
* Is available for clinical follow-up through Week 28 after enrollment.
* Has chronic HIV infection based on documentation from a primary care physician that the participant has HIV and is on antiretroviral therapy (ART).
* Is on a stable regimen of ART.
* Has at least 2 years of maintained HIV ribonucleic acid (RNA) < 50 copies/mL (or < lower limit of quantification [LLOQ] if the local laboratory assay's LLOQ is ≥50 copies/mL) prior to Screening and HIV RNA<50 at screening.
* Has CD4 cell count ≥350 cells/mm^3 at Screening.
* Is able to communicate effectively with the study investigator and other key personnel
* Has a primary care doctor for their medical management
* Is willing to donate blood for sample storage to be used for future research
* Female study participants with childbearing potential (defined below) and male study participants with female partners of childbearing potential must be willing to practice either:

  * Complete abstinence from sexual intercourse with a member of the opposite sex OR
  * Uses at least one form of effective contraception, in addition to correct use of either a male or female condom throughout dosing and for a defined period following the last dose (30 days for women, 14 days for men) of study medication

    * Definition of Childbearing Potential: For the purposes of this study, a female subject is considered of childbearing potential from menarche until becoming post-menopausal, unless permanently sterile or with medically documented ovarian failure. Women are considered to be in a post-menopausal state when they are ≥ 54 years of age with cessation of previously occurring menses for ≥ 12 months without an alternative cause. Permanent sterilization includes hysterectomy, bilateral oophorectomy, or bilateral salpingectomy in a female subject of any age.
* Agrees to adhere to Lifestyle Considerations throughout study duration

Exclusion Criteria:

* Has a current or prior history of any of the following:

  1. Clinically significant illness (other than HIV) or any other major medical disorder that may, in the opinion of the investigator, interfere with the participant treatment, assessment of compliance with the protocol; participants currently under evaluation for a clinically-significant illness (other than HIV) are also excluded
  2. Poor venous access interfering with required study blood collection
  3. Solid organ transplantation
  4. Significant pulmonary disease, significant cardiac disease, or porphyria
  5. Uncontrolled chronic hepatitis B infection (surface antigen positive with detectable HBV DNA as noted in participant's medical documentation from a treating physician)
  6. Chronic, current/active hepatitis C infection
  7. Unstable psychiatric disease. (Subjects with psychiatric illness that is well-controlled on a stable treatment regimen or currently not requiring medication may be included.)
  8. Any malignancy or its treatment that in the opinion of the Principal Investigator (PI) may cause ongoing interference with host immunity; subjects under evaluation for malignancy are not eligible.
* Has abnormal hematological and biochemical parameters at screening, unless the test has been repeated and at least one subsequent result is within the acceptable range prior to study drug administration, including:

  1. Neutrophil count <750 cells/mm^3
  2. Hemoglobin level <10 g/dL
  3. Platelet count ≤50,000 cells/mm^3
  4. Estimated glomerular filtration rate, calculated by the chronic kidney disease epidemiology collaboration formula: <30 mL/min/1.73 m^2
  5. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≥5 times upper limit of normal (ULN)
  6. Total bilirubin level ≥2.0 times ULN, except in subjects with Gilbert's syndrome or other clinical explanation at the discretion of the PI
  7. Albumin level <3 g/dL
* Has poorly controlled diabetes as indicated by a screening glycosylated hemoglobin (HbA1c) >10
* Has need for the use of the following medications from 21 days prior to the start of study drugs through the end of treatment:

  1. Hematologic stimulating agents, erythropoiesis stimulating agents (ESAs), granulocyte colony stimulating factor (GCSF), thrombopoeitin (TPO) mimetics
  2. Chronic systemic antineoplastic or immunomodulatory treatment including supraphysiologic doses of immunosuppressants such as corticosteroids (e.g., prednisone equivalent >10 mg/day for >2 weeks), azathioprine or monoclonal antibodies (e.g., infliximab)
  3. Investigational agents or devices for any indication
* Has hyperlipidemia (defined as an LDL ≥190 mg/dL), that is not being treated with 2018 ACC/AHA Cholesterol Clinical Practice guidelines (statins, Ezetimibe, PCSK9 inhibitors)
* Has a known history of cardiac arrhythmia or baseline ECG with arrhythmia including but not limited to atrial fibrillation (with or without rapid ventricular rate), supraventricular tachycardia or ventricular tachycardia.
* Has any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.
* Is a female who is breast-feeding or planning to become pregnant during the first 24 weeks after study drug administration.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Institute of Human Virology, University of Maryland Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Tian RR, Zhang MX, Zhang LT, Zhang P, Ma JP, Liu M, Devenport M, Zheng P, Zhang XL, Lian XD, Ye M, Zheng HY, Pang W, Zhang GH, Zhang LG, Liu Y, Zheng YT. CD24 and Fc fusion protein protects SIVmac239-infected Chinese rhesus macaque against progression to AIDS. Antiviral Res. 2018 Sep;157:9-17. doi: 10.1016/j.antiviral.2018.07.004. Epub 2018 Jul 3. PMID 29983395
- [Background] Tian RR, Zhang MX, Liu M, Fang X, Li D, Zhang L, Zheng P, Zheng YT, Liu Y. CD24Fc protects against viral pneumonia in simian immunodeficiency virus-infected Chinese rhesus monkeys. Cell Mol Immunol. 2020 Aug;17(8):887-888. doi: 10.1038/s41423-020-0452-5. Epub 2020 May 7. No abstract available. PMID 32382131
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 8 participants were randomized at 1 study site in the United States.
Groups:
- CD24Fc 240 mg: Participants received an intravenous infusion of 240 mg of CD24Fc on Days 0, 14, and 28.
Period: Overall Study
Arm/Group | CD24Fc 240 mg | Placebo
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CD24Fc 240 mg | Placebo | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.5 (1.73) | 58.8 (7.59) | 55.6 (6.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Low-Density Lipoprotein-Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] — LDL-C was measured in participant serum.
  mg/dL | 108.8 (22.38) | 116.0 (46.01) | 112.4 (33.72)
Serum Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Total cholesterol was measured in participant serum.
  mg/dL | 182.5 (40.17) | 190.0 (47.57) | 186.3 (40.96)
Serum High-Density Lipoprotein-Cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] — HDL-C was measured in participant serum.
  mg/dL | 52.0 (20.59) | 49.3 (8.18) | 50.6 (14.58)
Serum Triglycerides [Mean (Standard Deviation); unit: mg/dL] — Triglycerides were measured in participant serum.
  mg/dL | 121.5 (47.47) | 141.8 (68.01) | 131.6 (55.36)
Controlled Attenuation Parameter (CAP) [Mean (Standard Deviation); unit: Decibels/meter (dB/m)] — Controlled Attenuation Parameter (CAP) was measured using Transient Elastography of the Liver.
  Decibels/meter (dB/m) | 237.5 (115.07) | 215.5 (27.26) | 226.5 (78.30)
Liver Stiffness [Mean (Standard Deviation); unit: Kilopascal (kPa)] — Liver stiffness was measured using Transient Elastography of the liver.
  Kilopascal (kPa) | 5.65 (3.348) | 5.40 (1.699) | 5.53 (2.462)
Serum Leptin [Mean (Standard Deviation); unit: µg/L] — Leptin was measured in participant serum.
  µg/L | 27.65 (27.641) | 18.63 (30.388) | 23.14 (27.322)
Percent Glycated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage of Hemoglobin] — HbA1c was measured in participant blood.
  Percentage of Hemoglobin | 5.98 (0.918) | 5.55 (0.191) | 5.76 (0.655)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-Density Lipoprotein-Cholesterol (LDL-C)
Description: LDL-C was measured in participant serum. The percent change from baseline at Week 6 is presented.
Time Frame: Baseline and Week 6
Population: All randomized participants who received ≥1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | CD24Fc 240 mg | Placebo
Number analyzed (Participants) | 4 | 4
Percent Change | 6.24 (6.392) | 6.51 (19.690)

2. Primary Outcome: Number of Participants With ≥1 Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Any worsening of a preexisting condition which is temporally associated with the use of the study treatment is also considered an AE. The number of participants who experienced an AE is presented.
Time Frame: Up to approximately 28 weeks
Population: All randomized participants who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | CD24Fc 240 mg | Placebo
Number analyzed (Participants) | 4 | 4
Participants | 4 | 4

3. Primary Outcome: Number of Participants Who Withdrew From Study Treatment Due to an AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Any worsening of a preexisting condition which is temporally associated with the use of the study treatment is also considered an AE. The number of participants who withdrew from study treatment due to an AE is presented.
Time Frame: Up to approximately 4 weeks
Population: All randomized participants who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | CD24Fc 240 mg | Placebo
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

4. Secondary Outcome: Percent Change From Baseline in Total Cholesterol, High-Density Lipoprotein-Cholesterol (HDL-C), and Triglycerides
Description: Total cholesterol, HDL-C, and triglycerides were measured in participant serum. The percent change from baseline at Weeks 6 and 28 for these lipid panel results is presented.
Time Frame: Baseline, Week 6, and Week 28
Population: All randomized participants who received ≥1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | CD24Fc 240 mg | Placebo
Number analyzed (Participants) | 4 | 4
Percent Change
  Percent Change from Baseline in Total Cholesterol at Week 6 | 4.66 (5.850) | 1.53 (10.947)
  Percent Change from Baseline in HDL-C at Week 6 | 6.69 (12.250) | 0.88 (6.655)
  Percent Change from Baseline in Triglycerides at Week 6 | -8.42 (24.982) | -7.30 (23.607)
  Percent Change from Baseline in Total Cholesterol at Week 28 | 5.61 (21.672) | 2.40 (18.037)
  Percent Change from Baseline in HDL-C at Week 28 | 0.30 (0.610) | 3.20 (19.512)
  Percent Change from Baseline in Triglycerides at Week 28 | -2.77 (48.320) | -1.80 (46.310)

5. Secondary Outcome: Percent Change From Baseline in Cluster of Differentiation 4 (CD4)+ and Cluster of Differentiation 8 (CD8)+ T Cell Percentage
Description: The percent change from baseline in the percentage of T Cells in whole blood that are CD4+ and CD8+ at Weeks 6 and 28 was to be presented.
Time Frame: Baseline, Week 6, and Week 28
Population: The intended analysis population was all randomized participants who received ≥1 dose of study drug. Data for this outcome measure could not be collected because the laboratory was unable to run the assay. Therefore, no participants were analyzed.
Arm/Group | CD24Fc 240 mg | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percent Change From Baseline in Interferon (IFN)+ Peripheral Blood Mononuclear Cells (PBMCs)
Description: The percent change from baseline in the percentage of PBMCs that were INF+ at Weeks 6 and 28 was to be presented.
Time Frame: Baseline, Week 6, and Week 28
Population: as for outcome 5
Arm/Group | CD24Fc 240 mg | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percent Change From Baseline in Tumor Necrosis Factor (TNF)+ Peripheral Blood Mononuclear Cells (PBMCs)
Description: The percent change from baseline in the percentage of PBMCs that were TNF+ at Weeks 6 and 28 was to be presented.
Time Frame: Baseline, Week 6, and Week 28
Population: as for outcome 5
Arm/Group | CD24Fc 240 mg | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Percent Change From Baseline in Whole Blood Soluble Cluster of Differentiation 14 (sCD14) Concentration
Description: The percent change from baseline in sCD14 concentration in whole blood at Weeks 6 and 28 was to be presented.
Time Frame: Baseline, Week 6, and Week 28
Population: as for outcome 5
Arm/Group | CD24Fc 240 mg | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change From Baseline in Human Immunodeficiency Virus (HIV) Proviral Deoxyribonucleic Acid (DNA)
Description: Blood was collected at baseline, Week 6, and Week 28 for the determination of the number of copies of HIV proviral DNA in PBMCs. The change from baseline at Weeks 6 and 28 was to be presented.
Time Frame: Baseline, Week 6, and Week 28
Population: as for outcome 5
Arm/Group | CD24Fc 240 mg | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Percent Change From Baseline in Troponin I and Troponin T Serum Levels
Description: Troponin I and troponin T blood concentrations were to be measured. The percent change from baseline at Week 28 was to be presented.
Time Frame: Baseline and Week 28
Population: The intended analysis population was all randomized participants who received ≥1 dose of study drug. Results for baseline and/or Week 28 were not quantifiable for any participants, so the change from baseline analysis could not be performed and no participants were analyzed.
Arm/Group | CD24Fc 240 mg | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Percent Change From Baseline in Controlled Attenuation Parameter (CAP) as Determined by Transient Elastography of the Liver
Description: CAP is a measure related to hepatic steatosis. CAP was measured in decibels per meter (dB/m) at baseline and Week 28. The percent change is presented.
Time Frame: Baseline and Week 28
Population: All randomized participants who received ≥1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | CD24Fc 240 mg | Placebo
Number analyzed (Participants) | 4 | 4
Percent Change | 23.98 (34.167) | -5.86 (33.756)

12. Secondary Outcome: Percent Change From Baseline in Liver Stiffness as Determined by Transient Elastography of the Liver
Description: Liver stiffness is a measure related to hepatic fibrosis. Liver stiffness was measured in kilopascals (kPa) at baseline and Week 28. The percent change is presented.
Time Frame: Baseline and Week 28
Population: All randomized participants who received ≥1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | CD24Fc 240 mg | Placebo
Number analyzed (Participants) | 4 | 4
Percent Change | -0.81 (52.168) | 16.16 (27.449)

13. Secondary Outcome: Percent Change From Baseline in Leptin
Description: Leptin concentration was measured in participant serum. The percent change from baseline at Weeks 6 and 28 is presented.
Time Frame: Baseline, Week 6, and Week 28
Population: All randomized participants who received ≥1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | CD24Fc 240 mg | Placebo
Number analyzed (Participants) | 4 | 4
Percent Change
  Percent Change from Baseline at Week 6 | 46.72 (36.104) | 22.43 (73.205)
  Percent Change from Baseline at Week 28 | 83.03 (117.848) | 29.84 (84.316)

14. Secondary Outcome: Percent Change From Baseline in Glycated Hemoglobin (HbA1c)
Description: Glycated hemoglobin (HbA1c) is a blood marker used to report average blood glucose levels over prolonged periods of time. Percentage HbA1c is the ratio of glycated hemoglobin to total hemoglobin x 100. The percent change from baseline at Weeks 6 and 28 is presented.
Time Frame: Baseline, Week 6, and Week 28
Population: All randomized participants who received ≥1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | CD24Fc 240 mg | Placebo
Number analyzed (Participants) | 4 | 4
Percent Change
  Percent Change from Baseline at Week 6 | 0.69 (3.665) | -2.71 (1.070)
  Percent Change from Baseline at Week 28 | 4.65 (2.585) | 0.03 (2.557)

15. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of CD24Fc
Description: AUC was defined as the area of plasma concentration versus time curve from time zero to Week 28. Assessment of AUC was to be based on CD24Fc concentration measured in plasma samples collected at each study visit starting with Week 0.
Time Frame: Predose and 2 hours postdose at the Week 0, 2, and 4 visits; Any time during the Week 6, 16, and 28 visits.
Population: The intended analysis population was all randomized participants who received ≥1 dose of study drug. The estimated time to set up new validated assays exceeds the known stability of collected samples; therefore the samples will not be analyzed. Therefore, no participants were analyzed.
Arm/Group | CD24Fc 240 mg | Placebo
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Number of Participants With New Anti-Drug Antibodies
Description: Anti-CD24Fc antibodies were to be quantified in participant blood samples. The number of participants who demonstrated development of new anti-drug antibodies were to be presented.
Time Frame: Baseline, Week 6, and Week 28
Population: as for outcome 15
Arm/Group | CD24Fc 240 mg | Placebo
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Change From Baseline in Interluekin-6 (IL-6) Levels Following CD24Fc Treatment
Description: Levels of IL-6 were to be measured in participant blood samples collected at baseline and Week 28. The change from baseline in IL-6 levels were to be presented.
Time Frame: Baseline and Week 28
Population: The intended analysis population was all randomized participants who received ≥1 dose of study drug. No samples were collected for Week 28, so the change from baseline analysis could not be performed and no participants were analyzed.
Arm/Group | CD24Fc 240 mg | Placebo
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Change From Baseline in Apolipoprotein B (apoB) Levels
Description: Levels of apoB were measured in participant blood samples collected at baseline and Week 28. The change from baseline level is presented.
Time Frame: Baseline and Week 28
Population: All randomized participants who received ≥1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CD24Fc 240 mg | Placebo
Number analyzed (Participants) | 4 | 4
mg/dL
  Baseline | 109.0 (19.34) | 105.0 (29.31)
  Change from Baseline | -9.8 (14.75) | 6.5 (25.09)

19. Secondary Outcome: Change From Baseline in Lipoprotein(a) (Lp[a]) Levels
Description: Levels of Lp(a) were measured in participant blood samples collected at baseline and Week 28. The change from baseline level is presented.
Time Frame: Baseline and Week 28
Population: All randomized participants who received ≥1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CD24Fc 240 mg | Placebo
Number analyzed (Participants) | 4 | 4
mg/dL
  Baseline | 60.38 (39.443) | 301.45 (140.645)
  Change from Baseline | -15.03 (9.662) | 8.40 (70.528)

20. Secondary Outcome: Change From Baseline in Urine Albumin:Creatinine Ratio
Description: The ratio between levels of albumin and creatine was measured in participant urine at baseline and Week 28. The change from baseline in the ratio is presented.
Time Frame: Baseline and Week 28
Population: All randomized participants who received ≥1 dose of study drug and had data available for the specified time point.
Measure: Mean (Standard Deviation); unit: Ratio (g Albumin/mol Creatinine)
Arm/Group | CD24Fc 240 mg | Placebo
Number analyzed (Participants) | 3 | 3
Ratio (g Albumin/mol Creatinine)
  Baseline | 6.0 (2.65) | 796.3 (1322.45)
  Change from Baseline | 0.5 (0.71) | -357.0 (434.16)

21. Other Pre Specified Outcome: Change From Baseline in Aortic F-fluorodeoxyglucose (FDG) Uptake
Description: Arterial FDG uptake is used to evaluate arterial inflammation. Arterial FDG uptake was to be measured by positron emission tomography-computed tomography (PET/CT) scan at Baseline and Week 24 in the aortic root and the same superior vena cava, then reported as the aortic uptake value divided by the superior vena cava uptake value, the target-to-background ratio (TBR). The change from baseline at Week 24 was to be presented.
Time Frame: Baseline and Week 24
Population: The intended analysis population was the first 12 randomized participants who received ≥1 dose of study drug, had LDL levels greater than 125 mg/dL, and volunteered for this optional measurement. No participants volunteered for the PET/CT scans required for this outcome measure. Therefore, no participants were analyzed.
Arm/Group | CD24Fc 240 mg | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for up to approximately 28 weeks. All-Cause Mortality was monitored for up to approximately 36 weeks.
Description: All-Cause Mortality includes all randomized participants. Adverse Events include participants who received ≥1 dose of study treatment.
Arm/Group | CD24Fc 240 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD24Fc 240 mg (N=4) | Placebo (N=4)
Glomerular filtration rate decreased (Investigations) | 3 (4) | 2 (4)
Blood albumin decreased (Investigations) | 2 (2) | 0 (0)
Blood cholesterol increased (Investigations) | 2 (2) | 2 (6)
Blood glucose increased (Investigations) | 2 (4) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 2 (2)
Prothrombin time prolonged (Investigations) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (2)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (2)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 1 (1)
Coronavirus test positive (Investigations) | 0 (0) | 1 (1)
Low density lipoprotein increased (Investigations) | 0 (0) | 2 (6)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 4 (18) | 4 (17)
Sinus bradycardia (Cardiac disorders) | 2 (3) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any reports, papers, and/or presentations must be reviewed and approved by the sponsor prior to submitting for publication. All publications relating to the study will comply with the guidelines set forth by the Uniform Requirements for Manuscripts Submitted to Biomedical Journals drawn up by the International Committee of Medical Journal Editors.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/41/NCT03960541/Prot_SAP_000.pdf